CLINICAL TRIAL: NCT05659849
Title: Effectiveness of Manual Therapy VS Conventional Physical Therapy With Neuromuscular Training in the Management of Knee Osteoarthritis
Brief Title: Effectiveness of Manual Therapy and Neuromuscular Training in the Management of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tabuk (Other)
Responsible Party: Principal Investigator, Shahul Hameed Pakkir Mohamed, ASSOCIATE PROFESSOR, University of Tabuk
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UT-217-68-2022
Record Dates: First submitted 2022-12-12; First posted 2022-12-21 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee; Osteoarthritis; Manual therapy; TENS; Neuromuscular training
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy with Neuromuscular training (Experimental): Manual physical therapy is intended to improve musculoskeletal function and pain by addressing impaired kinematics of the joint. Passive Joint Mobilization (PJM) was applied to knee distraction and dorsal glides, ventral glides, and patellar glides in all directions, which were applied at a rate of two to three oscillations per second for 1-2 min. Each direction was repeated three to six times.
  Neuromuscular training (NEMEX-TJR training program):
  (2 times per week for 6 weeks) The neuromuscular training program consists of 3 parts: warming up, a circuit program, and cooling down. The program is performed twice a week for 6 weeks, with each session lasts for 60 minutes.
  Interventions: Other: Manual therapy techniques
- Conventional physical therapy with Neuromuscular training (Experimental): Physical therapists use a variety of transcutaneous electrical nerve stimulation (TENS) applications to reduce or alleviate pain for individuals with Knee OA. TENS (symmetrical biphasic waveform, frequency 32-50 Hz, pulse width 80 microseconds) for the same amount of time and the same number of days. The TENS electrodes were applied on the medial and lateral superior, as well as the medial and lateral inferior, borders of the patella. Care was taken not to place TENS electrodes on the quadriceps muscles or muscles of the anterior leg.
  Neuromuscular training (NEMEX-TJR training program):
  (2 times per week for 6 weeks) The neuromuscular training program consists of 3 parts: warming up, a circuit program, and cooling down. The program is performed twice a week for 6 weeks, with each session lasts for 60 minutes.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Other: Manual therapy techniques — Passive joint mobilization techniques are applied to the affected knee joint. For the first week (three sessions), the joint mobilization exercises included grade I or II rhythmic oscillations. During the following weeks, grade III or IV oscillation techniques were applied, depending on the level of tolerance and pain of each patient. In knee distraction, the patients are in a prone position with 50° knee flexion, and the physical therapist applies the techniques. The dorsal and ventral glides was performed with the patient in a supine position.
  Arms: Manual therapy with Neuromuscular training
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — Transcutaneous electrical nerve stimulation (TENS) therapy treats pain using low-voltage electric currents. A small device administers the electrical current to or near nerves. TENS treatment inhibits or changes pain perception.
  Arms: Conventional physical therapy with Neuromuscular training

SUMMARY:
The purpose of the study is to compare the short-term effectiveness of manual therapy with neuromuscular training and conventional physical therapy with neuromuscular training in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a major public health problem, characterized by progressive degeneration and loss of articular cartilage, resulting in pain, limitation of movement, imbalance, functional disability, and diminished patient quality of life. Regular participation in physical activity has been recognized for several years as being beneficial in the management of knee OA. The role and effectiveness of manual therapy techniques and conventional physical therapy are evident from the existing literature, but no comparison was found for the combination of neuromuscular training (NMT) in patients with knee OA. Thus, the aim of this study is to compare the short-term effectiveness of manual therapy (MT) versus conventional physical therapy (CPT) with NMT in the management of knee OA after six weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Complaining of knee pain that has lasted longer than 3 months.
* Pain level that is medium (pain score greater than or equal to 4).
* No knee injuries.
* Treatment not received in another physical therapy clinic in the past three months.
* Painful range of motion in the knee.

Exclusion Criteria:

* History of knee surgery
* A systemic arthritic condition
* Any other muscular, joint, or neurological condition affecting lower limb function.
* Received physical therapy or an intra-articular injection in the knee within the past 3 months.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 6 weeks
  The average pain intensity over the last week at the time of testing was measured on a numerical pain rating scale, where 0 represented no pain and 10 represented the worst pain possible.
Goniometric measurement for ROM | 6 weeks
  To check the range of motion (ROM) of the knee joint, the joint will be extended as far as it can go while the person is lying on their back three times. The angle at the maximum flexion position was measured with a goniometer, and the average angle was recorded.
Western Ontario and Mc Master Osteoarthritis Index (WOMAC) | 6 weeks
  It is a questionnaire for the evaluation of treatment results in patients with lower extremity osteoarthritis, and it divides difficulties in daily living into scales. WOMAC scores are recorded on a five-point Likert scale of 0-4, where 0 = no pain or limitation, 1 = mild pain or limitation, 2 = moderate pain or limitation, 3 = severe pain or limitation, and 4 = extreme pain or limitation. Maximum scores for pain, stiffness and physical functions were 20, 8, and 68, respectively, with total scores of 96 indicating greater disease severities.
Short-Form Health Survey (SF-36) | 6 weeks
  This instrument consists of 36 items, grouped into eight domains: functional capacity, physical aspects, pain, general health, vitality, social aspects, emotional aspects, and mental health. A measurement scale with values ranging from 0 (the worst health status) to 100 (the best health status) was used to give each subject and each of the eight dimensions a score.
Single-leg stance time test | 6 weeks
  This test has been used to assess static standing balance in individuals with knee OA. The single-leg stance test was measured by recording the time in seconds (30s maximum) while participants are asked to balance on one leg while keeping their hands on their hips. The test starts when the free foot lifts off the ground and is stopped if: (1) the swing limb touches the ground; (2) the stance foot moves on the floor; (3) the swing foot touches the tested limb; or (4) the hands move away from the hips.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tabuk, Tabuk, North West, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No